CLINICAL TRIAL: NCT07076979
Title: Development and Validation of Metabolic Biomarkers for Early Diagnosis, Prognosis, and Recurrence of Gastric：MetBio-GC
Brief Title: Development and Validation of Metabolic Biomarkers for Early Diagnosis, Prognosis, and Recurrence of Gastric Cancer：MetBio-GC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: MetBio-GC
Record Dates: First submitted 2025-07-08; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Metabolic marker; Prognosis; Early diagnosis
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Peripheral blood samples and tumor tissue samples are collected accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline: This group recruits healthy individuals which is intended to establish a metabolic biomarker baseline
- GC: Gastric cancer group, which is study of interest

SUMMARY:
This prospective clinical observational study aims to construct a metabolite database specifically for gastric cancer patients using metabolomics technology. It seeks to develop and validate metabolic biomarkers for early diagnosis, prognosis, and prediction of recurrence and metastasis in gastric cancer, thereby a establishing safe, convenient, and highly sensitive method for early screening and prognostic prediction.

ELIGIBILITY:
Inclusion Criteria:

* **Healthy Controls:**

  1. Age > 18 years;
  2. Signed informed consent and willingness to participate in the project.

**Gastric Cancer:**

1. Age ≥ 18 years;
2. Performance status (ECOG) score ≤ 1;
3. Histopathologically confirmed gastric adenocarcinoma;
4. No family history of hereditary cancer;
5. No prior anti-tumor treatment;
6. Availability of primary tumor tissue from surgery or biopsy that meets submission requirements;
7. Availability of peripheral blood samples that meet submission requirements;
8. Willingness and ability to sign the informed consent form to participate in the study.

Exclusion Criteria:

* **Healthy Controls:**

  1. Individuals at high risk for hereditary colorectal adenocarcinoma, including family members of the following diseases: family history of gastrointestinal tumors, familial adenomatous polyposis (FAP), hereditary nonpolyposis colorectal cancer (HNPCC/LS), and Peutz-Jeghers syndrome (P-J syndrome);
  2. History of chronic metabolic or inflammatory diseases that are difficult to control, such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease;
  3. Known history of other malignancies that have progressed or required treatment within the past 5 years, except for skin basal cell carcinoma and squamous cell carcinoma that have been cured;
  4. History of oral or intravenous use of broad-spectrum antibiotics and probiotics within the past month;
  5. Regular use of immunosuppressive drugs within the past 6 months;
  6. Long-term use of other medications that may affect metabolism, such as hormones;
  7. Inability or unwillingness to cooperate with follow-up visits and related examinations;
  8. Inability to eat normally or requiring medications or enemas for bowel movements;
  9. Presence of psychiatric disorders or other severe cardiovascular diseases;
  10. Pregnant, breastfeeding, or planning to become pregnant within the next year;
  11. Currently participating in an interventional clinical study or receiving study treatment that may influence the patient's treatment decision.

**Gastric Cancer:**

1. Currently participating in an interventional clinical study or receiving study treatment that may influence the patient's treatment decision;
2. Known history of other malignancies that have progressed or required treatment within the past 5 years, except for skin basal cell carcinoma and squamous cell carcinoma that have been cured;
3. History of chronic metabolic or inflammatory diseases that are difficult to control, such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease;
4. Presence of poorly controlled chronic comorbidities that may affect prognosis;
5. Presence of psychiatric disorders or other severe cardiovascular diseases;
6. Pregnant, breastfeeding, or planning to become pregnant within the next year;
7. Long-term use of medications that may affect metabolism, such as hormones, immunosuppressants, antibiotics, etc.;
8. Any severe and/or uncontrolled medical conditions, as judged by the investigator, that may affect the patient's ability to participate in the study or interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  The time from the start of treatment to death due to any cause.
Disease-Free Survival | 3 years
  Disease-Free Survival (DFS) refers to the length of time after primary treatment for a disease during which the patient remains free of certain signs or symptoms of the disease. It is typically measured from the start of treatment until the first recurrence or relapse of the disease.

SECONDARY OUTCOMES:
Hazard Ratio | 3 years
  The hazard ratio is a measure of the relative risk of an event occurring in one group compared to another group. It is used to quantify the difference in the rate at which events occur between two groups, typically a treatment group and a control group.
Positive Predictive Value | 3 years
  The Positive Predictive Value (PPV) indicates how likely it is that a person actually has the disease if the test result is positive.
Negative Predictive Value | 3 years
  The Negative Predictive Value (NPV) indicates how likely it is that a person does not have the disease if the test result is negative.
Assessment of Important Metabolic Biomarkers | 3 years
  This outcome measure is intended to identify important metabolic biomarkers that are highly statistically associated with the prognosis of gastric cancer, such as OS, DFS, etc., given different time frames.
Recurrence Rate | 3 years
Cancer-Related Mortality | 3 years
Time to Recurrence and Metastasis and Specific Sites | 3 years
Distant Metastasis Rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital Shanghai Jiaotong University, School of Medicine , Shanghai, Shanghai 200025, Shanghai, China

IPD SHARING:
Plan to Share IPD: No